CLINICAL TRIAL: NCT05012267
Title: OptiMal pronE Position LEnghT in Patients With acuTE Respiratory Distress Syndrome Due to COVID-19.
Brief Title: Duration of Prone Position in the Severe Acute Respiratory Syndrome Coronavirus 2 (COVID-19).
Acronym: OmeLEtte
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ignacio Saez de la Fuente (Other)
Responsible Party: Sponsor-Investigator, Ignacio Saez de la Fuente, Ignacio Saez de la Fuente, MD, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMELETTE
Record Dates: First submitted 2021-08-11; First posted 2021-08-19 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Ards
Keywords: prone position; mechanical ventilation; oxygenation
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): 48 hours of PP
- Experimental group (Experimental): Anytime from 16 hours when PaO2/FiO2 ≥ 150 mmHg with a FiO2 < 60%
  Interventions: Other: 16-hour PP

INTERVENTIONS:
Other: 16-hour PP — PP according to previous study
  Arms: Experimental group

SUMMARY:
The OMELETTE study is a randomised, controlled, unicentric, open-label study to prove the noninferiority of reduced prone position (PP) sessions (more tan 16 hours) versus prolonged PP (48 hours).

DETAILED DESCRIPTION:
This is a non-comercial, investigator-driven clinical study developed in a single critical care unit.

The study is coordinated by the main investigator from Hospital Universitario 12 de Octubre in Madrid; The sponsorship is performed by Dr. Ignacio Sáez (Hospital Universitario 12 de Octubre).

The study was planned according to the Good Clinical Practices. Omelette study has been approved by the Ethics Committee. All participating Patients must give informed consent before any study procedure occur.

ELIGIBILITY:
Inclusion Criteria:

* Patient above 18 year-old.
* Diagnosis of severe ARDS due to COVID-19 under invasive mechanical ventilation,
* Meet criteria for PP: PaO2/FiO2 < 150 millimeters of mercury column (mmHg), PEEP ≥ 5 Centimeters of Water (cmH2O), FiO2 ≥ 60.

Exclusion Criteria:

* No consent for the study.
* PP contraindicated (( elevated intracranial pressure, massive hemoptysis, recent tracheal surgery or sternotomy, unstable hemodynamic status, recent pacemaker implantation, severe facial laceration, open abdominal wound, spine, femur or pelvis fracture or pregnancy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Ventilator-free days at 28 days | 28 days
  Number of days from successfully weaning to day 28
Ventilator-free days at 60 days | 60 days
  Number of days from successfully weaning to day 60

SECONDARY OUTCOMES:
Survival | 60 days
  Mortality during ICU or hospital admission
ICU and Hospital stay | Hospital admission
  Days of stay
Evolution of respiratory parameters | ICU admission
  Measurement of mechanical ventilation parameters.
PP complications | ICU admission
  Proportion of Patients experiencing accidental removal of catheters, endotracheal tube obstruction or any serious adverse event.

OTHER OUTCOMES:
Enteral nutrition administration | ICU admission
  Nutritional intake.

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Sáez, MD, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang C, Horby PW, Hayden FG, Gao GF. A novel coronavirus outbreak of global health concern. Lancet. 2020 Feb 15;395(10223):470-473. doi: 10.1016/S0140-6736(20)30185-9. Epub 2020 Jan 24. No abstract available. PMID 31986257
- [Background] Ramirez P, Gordon M, Martin-Cerezuela M, Villarreal E, Sancho E, Padros M, Frasquet J, Leyva G, Molina I, Barrios M, Gimeno S, Castellanos A. Acute respiratory distress syndrome due to COVID-19. Clinical and prognostic features from a medical Critical Care Unit in Valencia, Spain. Med Intensiva (Engl Ed). 2021 Jan-Feb;45(1):27-34. doi: 10.1016/j.medin.2020.06.015. Epub 2020 Jul 11. PMID 32919796
- [Background] Mora-Arteaga JA, Bernal-Ramirez OJ, Rodriguez SJ. The effects of prone position ventilation in patients with acute respiratory distress syndrome. A systematic review and metaanalysis. Med Intensiva. 2015 Aug-Sep;39(6):359-72. doi: 10.1016/j.medin.2014.11.003. Epub 2015 Jan 17. English, Spanish. PMID 25599942
- [Background] Gattinoni L, Tognoni G, Pesenti A, Taccone P, Mascheroni D, Labarta V, Malacrida R, Di Giulio P, Fumagalli R, Pelosi P, Brazzi L, Latini R; Prone-Supine Study Group. Effect of prone positioning on the survival of patients with acute respiratory failure. N Engl J Med. 2001 Aug 23;345(8):568-73. doi: 10.1056/NEJMoa010043. PMID 11529210
- [Background] Mentzelopoulos SD, Roussos C, Zakynthinos SG. Prone position reduces lung stress and strain in severe acute respiratory distress syndrome. Eur Respir J. 2005 Mar;25(3):534-44. doi: 10.1183/09031936.05.00105804. PMID 15738300
- [Background] Galiatsou E, Kostanti E, Svarna E, Kitsakos A, Koulouras V, Efremidis SC, Nakos G. Prone position augments recruitment and prevents alveolar overinflation in acute lung injury. Am J Respir Crit Care Med. 2006 Jul 15;174(2):187-97. doi: 10.1164/rccm.200506-899OC. Epub 2006 Apr 27. PMID 16645177
- [Background] Guerin C, Gaillard S, Lemasson S, Ayzac L, Girard R, Beuret P, Palmier B, Le QV, Sirodot M, Rosselli S, Cadiergue V, Sainty JM, Barbe P, Combourieu E, Debatty D, Rouffineau J, Ezingeard E, Millet O, Guelon D, Rodriguez L, Martin O, Renault A, Sibille JP, Kaidomar M. Effects of systematic prone positioning in hypoxemic acute respiratory failure: a randomized controlled trial. JAMA. 2004 Nov 17;292(19):2379-87. doi: 10.1001/jama.292.19.2379. PMID 15547166
- [Background] Hermosilla J, Aguayo M, Ferreira L. [Total duration of ventilation in the prone position in patients with acute respiratory distress syndrome]. Med Intensiva. 2016 Jan-Feb;40(1):71. doi: 10.1016/j.medin.2015.09.006. Epub 2015 Nov 14. No abstract available. Spanish. PMID 26585675
- [Result] Mancebo J, Fernandez R, Blanch L, Rialp G, Gordo F, Ferrer M, Rodriguez F, Garro P, Ricart P, Vallverdu I, Gich I, Castano J, Saura P, Dominguez G, Bonet A, Albert RK. A multicenter trial of prolonged prone ventilation in severe acute respiratory distress syndrome. Am J Respir Crit Care Med. 2006 Jun 1;173(11):1233-9. doi: 10.1164/rccm.200503-353OC. Epub 2006 Mar 23. PMID 16556697
- [Result] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Result] Saez de la Fuente I, Saez de la Fuente J, Quintana Estelles MD, Garcia Gigorro R, Terceros Almanza LJ, Sanchez Izquierdo JA, Montejo Gonzalez JC. Enteral Nutrition in Patients Receiving Mechanical Ventilation in a Prone Position. JPEN J Parenter Enteral Nutr. 2016 Feb;40(2):250-5. doi: 10.1177/0148607114553232. Epub 2014 Oct 1. PMID 25274497
- [Result] Romero CM, Cornejo RA, Galvez LR, Llanos OP, Tobar EA, Berasain MA, Arellano DH, Larrondo JF, Castro JS. Extended prone position ventilation in severe acute respiratory distress syndrome: a pilot feasibility study. J Crit Care. 2009 Mar;24(1):81-8. doi: 10.1016/j.jcrc.2008.02.005. Epub 2008 May 14. PMID 19272543
- [Result] Concha P, Treso-Geira M, Esteve-Sala C, Prades-Berengue C, Domingo-Marco J, Roche-Campo F. Invasive mechanical ventilation and prolonged prone position during the COVID-19 pandemic. Med Intensiva (Engl Ed). 2021 Jan 16;46(3):161-3. doi: 10.1016/j.medin.2021.01.001. Online ahead of print. No abstract available. English, Spanish. PMID 33551113
- [Result] Jochmans S, Mazerand S, Chelly J, Pourcine F, Sy O, Thieulot-Rolin N, Ellrodt O, Mercier Des Rochettes E, Michaud G, Serbource-Goguel J, Vinsonneau C, Vong LVP, Monchi M. Duration of prone position sessions: a prospective cohort study. Ann Intensive Care. 2020 May 24;10(1):66. doi: 10.1186/s13613-020-00683-7. PMID 32449068